CLINICAL TRIAL: NCT01248767
Title: A Prospective Clinical Study of a Cohort of Pathological Patients Seeking Treatment for a Behavioral Addiction in the University Hospital of Nantes
Brief Title: A Prospective Clinical Study of a Cohort of Patients Seeking Treatment for a Behavioral Addiction
Acronym: EVALADD
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0004
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Behavioral Addictions
Keywords: cohort; cognitive distortions; impulsivity; psychiatric comorbidities; addiction; gambling disorder; sexual addiction; videogame disorder; food addiction; eating disorders; compulsive buying; behavioral addictions
MeSH Terms: conditions — Impulsive Behavior; Behavior, Addictive; Gambling; Compulsive Sexual Behavior Disorder; Food Addiction; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This research aims to provide a better understanding of the factors associated with the evolution of behavioral addictions, and compliance with care. The investigators thus aim to follow patients with several types of behavioral addictions, based on addictive, sociodemographic, clinical and endophenotypical characteristics, as well as their care adhesion.

ELIGIBILITY:
Inclusion Criteria :

- All consecutive patients seeking treatment at the University Hospital of Nantes for a behavioral addiction and age over 15 will be allowed to participate to the study.

Exclusion Criteria :

* Cognitive impairment incompatible with the assessment
* Difficulty for writing or reading the French language, incompatible with the assessement
* Gardianship

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking treatment for a behavioral addiction
Sampling Method: Non-Probability Sample
Enrollment: 2720 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Evolution of behavioral addictions | 8 years
  Understand what determines the evolution of behavioral addictions and compliance with care. Study the outcome of patients with behavioral addictions, both in terms of the evolution of of the addictive pathology and associated clinical and endophenotypic characteristics, as well as adherence to care.

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL-BRONNEC, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Challet-Bouju G, Caillon J, Leboucher J, Thiabaud E, Saillard A, Balem M, Grall-Bronnec M. Impact of Gambling on the Internet on Middle-Term and Long-Term Recovery from Gambling Disorder: A 2-Year Longitudinal Study. J Gambl Stud. 2025 Jun;41(2):567-592. doi: 10.1007/s10899-024-10328-0. Epub 2024 Sep 10. PMID 39254777